CLINICAL TRIAL: NCT04812132
Title: A Multicentre Randomized Controlled Trial Comparing Outcome of Laparoscopic One-anastomosis Gastric Bypass and Laparoscopic Long Biliopancreatic Limb Roux Gastric Bypass for Treatment of Morbid Obesity.
Brief Title: RCT Comparing OAGB and Long Limb Roux Gastric Bypass
Acronym: OAGBvsLLbypass
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tartu University Hospital (Other)
Collaborators: North Estonia Medical Centre (Other); Fertilitas (private clinic) (Unknown)
Responsible Party: Principal Investigator, Eva-Maria Kikkas, Doctor and Teaching staff, Tartu University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TartuUH
Record Dates: First submitted 2021-02-27; First posted 2021-03-23 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Obesity
Keywords: OAGB; Long biliary limb Roux gastric bypass; Metabolic surgery; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Women (Active Comparator)
  Interventions: Procedure: One-anastomosis gastric bypass; Procedure: Long biliary limb Roux gastric bypass
- Men (Active Comparator)
  Interventions: Procedure: One-anastomosis gastric bypass; Procedure: Long biliary limb Roux gastric bypass

INTERVENTIONS:
Procedure: One-anastomosis gastric bypass — One group is planned to have one-anastomosis gastric bypass (also known as mini-bypass)
Procedure: Long biliary limb Roux gastric bypass — Other group is planned to receive a long biliary limb Roux gastric bypass

SUMMARY:
A prospective multicenter randomized controlled trial to compare the outcomes of one-anastomosis gastric bypass to long biliary limb Roux gastric bypass.

We plan to enroll up to 500 patients from three different clinics in Estonia. Outcomes are excess weight loss %, impact on type 2 diabetes, hypertension, hyperlipidemia and obstructive sleep apnea.

Other outcomes are nutritional deficiencies, occurrence of reflux disease and impact on quality of life.

There are planned outpatient visits 1, 5 and 10 years after the surgery to measure the impacts.

There are a lot of studies comparing OAGB to standard Roux gastric bypass but non comparing it to long biliary limb gastric bypass.

ELIGIBILITY:
Inclusion Criteria:

* BMI over 35 and obesity related disease
* BMI over 40
* age between 18-60 years
* agrees to participate in the study

Exclusion Criteria:

* age under 18 years or over 60 years
* abundant adhesions discovered during the surgery
* active upper gastrointestinal ulcer disease
* prior bariatric surgery
* active symptomatic reflux disease
* active psychiatric disease (eg psychosis)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 500 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2031-12-31 (Estimated); Study Completion 2036-12-31 (Estimated)

PRIMARY OUTCOMES:
Excess weight loss % | 10 years
  Calculated loss of the excess weight
Impact on type 2 diabetes mellitus | 10 years
  Outcome of type 2 diabetes mellitus after the surgery, measured in change in HbA1c %
Impact on type 2 diabetes mellitus | 10 years
  Outcome of type 2 diabetes mellitus after the surgery, measured in usage of medication (same dosage, decreased dosage, insulin to peroral, ended all medication)
Impact on hypertensive disease | 10 years
  Outcome of hypertensive disease after the surgery; measured in antihypertensive drug usage (same, decrease, ended)
Impact on total cholesterol | 10 years
  Outcome of hyperlipidemias after the surgery, measured in change in levels of total cholesterol (mmol/L).
Impact on hyperlipidemia | 10 years
  Outcome of hyperlipidemias after the surgery, measured in change in levels of HDL (mmol/L)
Impact on hyperlipidemia | 10 years
  Outcome of hyperlipidemias after the surgery, measured in change in levels of LDL (mmol/L)
Impact on hyperlipidemia | 10 years
  Outcome of hyperlipidemias after the surgery, measured in change in levels of triglycerides (mmol/L)
Impact on hyperlipidemias | 10 years
  Outcome of hyperlipidemias after the surgery, measured in change in levels of total cholesterol, HDL,LDL and triglycerides

SECONDARY OUTCOMES:
Nutritional deficiencies: anemia | 10 years
  % of subjects having hemoglobin below sex adjusted reference (g/L) and ferritin below sex adjusted references (ug/L)
Nutritional deficiencies | 10 years
  Occurrence of B12 deficiency, measured in % of subjects with vitamin B12 below reference (measures in pmol/L)
GERD | 10 years
  % of subjects reporting reflux disease symptoms and/or PPI usage after the surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Tartu University Hospital, Tartu, Estonia

IPD SHARING:
Plan to Share IPD: No